CLINICAL TRIAL: NCT03938402
Title: Intraocular Pressure and Optic Nerve Sheath Diameter Changes at Different Positive End-expiratory Pressure Applications in Laparotomic Surgery
Brief Title: Intraocular Pressure and Optic Nerve Sheath Diameter Changes at Different PEEP Levels
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: As a result of COVID-19 pandemics
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ruslan Abdullayev, Assist. Prof., Marmara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 09.2019.378
Record Dates: First submitted 2019-04-27; First posted 2019-05-06 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Intraocular Pressure; Intracranial Pressure; Positive End-expiratory Pressure
Keywords: Intraocular pressure; Optic nerve sheath diameter; Positive end-expiratory pressure
MeSH Terms: interventions — Positive-Pressure Respiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PEEP 5 (Experimental)
  Interventions: Other: Positive end-expiratory pressure
- PEEP 10 (Experimental)
  Interventions: Other: Positive end-expiratory pressure
- PEEP 15 (Experimental)
  Interventions: Other: Positive end-expiratory pressure

INTERVENTIONS:
Other: Positive end-expiratory pressure — Different levels of positive end-expiratory pressure (i.e., 5, 10 and 15 cm H2O) will be applied to the groups.

SUMMARY:
Positive end-expiratory pressure (PEEP) is sometimes used during perioperative period, as it has favourable effects on lung mechanics. Unfortunately, it has some negative effects on the patients, like increased intraabdominal, intrathoracic, intracranial and intraocular pressures. In this study the investigators aimed to investigate the effects of different PEEP levels on the patients' intraocular and intracranial pressures. Intraocular pressure will be measured by ocular tonometry, and intracranial pressure will be estimated by optic nerve sheath diameter measurement. The measurements will be performed in the operating room in the patients undergoing laparotomic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparotomy for gastrointestinal surgery
* American Society of Anesthesiologists (ASA) 1 or 2 physical status
* Elective surgery

Exclusion Criteria:

* Patients with glaucoma
* ASA 3 or over physical status
* Emergency surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in intraocular pressure | Throughout the operation (usually about 1.5 hours).
  The physiological value for intraocular pressure is 10-20 mm Hg. Changes in intraocular pressure will be observed throughout the surgery, as will its relationship with the positive end-expiratory pressure application.
Changes in optic nerve sheath diameter | Throughout the operation (usually about 1.5 hours).
  Changes in optic nerve sheath diameter will be observed throughout the surgery, as will its relationship with the positive end-expiratory pressure application.

CONTACTS AND LOCATIONS:
Overall Officials: Ruslan Abdullayev, Principal Investigator — Marmara University School of Medicine, Dep of Anesthesiology and Reanimation
Locations (1):
- Marmara University School of Medicine, Istanbul, Pendik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No